CLINICAL TRIAL: NCT06026085
Title: A Prospective, Single-Center, Single-Blind, Randomized Split-Face Controlled Clinical Study to Evaluate the Efficacy and Satisfaction of the Skinceuticals Skin Care Product (CE FERULIC) for Skin Repair Post Fraxel Laser Treatment in Real World Clinical Practice
Brief Title: A Clinical Study to Evaluate the Efficacy and Satisfaction of the Skinceuticals Skin Care Product (CE FERULIC) for Skin Repair Post Fraxel Laser Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DeYi Aesthetic Medical Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKCFRX002
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Photo-damaging
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CE FERULIC (Experimental): fraxel laser therapy combined with Skinceuticals skin care product(CE FERULIC) and routine sun protection
  Interventions: Other: Skinceuticals skin care product(CE); Other: fraxel laser therapy
- 0.9% normal saline (Placebo Comparator): fraxel laser therapy combined with 0.9% normal saline and routine sun protection
  Interventions: Other: fraxel laser therapy; Other: 0.9% normal saline

INTERVENTIONS:
Other: Skinceuticals skin care product(CE) — Skinceuticals skin care product(CE FERULIC)+routine sun protection
  Arms: CE FERULIC
Other: fraxel laser therapy — Fraxel DUAL 1550/1927 Laser System
Other: 0.9% normal saline — 0.9% normal saline+routine sun protection
  Arms: 0.9% normal saline

SUMMARY:
A Prospective, Single-center, Single-blind, Randomized split-face, controlled trial will be conducted. The goal of this clinical trial is to evaluate the efficacy and satisfaction of the Skinceuticals skin care product (CE) for skin repair following fraxel laser treatment and explore the medical value of fraxel laser therapy combined with Skinceuticals skin care product

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 18-65 years (inclusive);
2. Subjects with Fitzpatrick skin type II-IV;
3. Subjects with mild to moderate facial photoaging lesions, including melasma, acne scars, fine skin lines, enlarged pores, and dark photoaging problems
4. Subjects with consistent facial skin status on both sides and planned to receive fraxel laser treatment;
5. Subjects are willing to follow the requirements of the study protocol and complete the corresponding procedures;
6. Subjects understand the nature of the study and sign the informed consent form (ICF)

Exclusion Criteria:

1. Subjects with photosensitive skin or photosensitization-related diseases;
2. Subjects with a history of skin pigmentation, such as pigmentation caused by sex hormone factors (pregnancy, oral contraceptives);
3. Subjects with hypertrophic scar or scar constitution;
4. Subjects with autoimmune diseases, endocrine diseases or liver diseases that may lead to skin color changes;
5. Subjects who have received steroid/phototoxic drugs or laser treatment on the face within 3 months before enrollment;
6. Subjects with a history of sun exposure within 2 weeks prior to enrollment;
7. Subjects who are known to be contraindicated to fraxel laser therapy or CE (or allergic to other skin care components);
8. Subjects with known infection and inflammation in the intended treatment site;
9. Female subjects who are pregnant, lactating or plan to become pregnant;
10. Subjects who plan to use other drugs affecting skin color or intend to undergo other laser therapy and sunbathing during the treatment;
11. Subjects who are participating in other drug or medical device clinical trials;
12. Other subjects who are not suitable for this study as assessed by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in erythema score | at day 7 post-procedure
  Scoring criteria: 0 (no erythema), 1 (mild erythema), 2 (moderate erythema), and 3 (severe erythema)

SECONDARY OUTCOMES:
Change from baseline in erythema score | days 1, 3 post-procedure
  Scoring criteria: 0 (no erythema), 1 (mild erythema), 2 (moderate erythema), and 3 (severe erythema)
Change from baseline in edema score | days 1, 3,7 post-procedure
  Score 0 - no edema, score 1 - mild edema, score 2 - moderate edema, score 3 - severe edema
Change from baseline in Erythema Index (EI) | days 1, 3,7 post-procedure
  EI values were measured on both sides of their faces with a multifunctional skin tester MPA20 (Courage Khazaka, Germany) + Mexameter MX18 probe
Change from baseline in melanin index(MI) | days 1, 3,7 post-procedure
  MI values were measured on both sides of their faces with a multifunctional skin tester MPA20 (Courage Khazaka, Germany) + Mexameter MX18 probe
Change from baseline in stratum corneum water content | days 1, 3,7 post-procedure
Change from baseline in transepidermal water loss | days 1, 3,7 post-procedure
Change from baseline in sebum rate | days 1, 3,7 post-procedure
Subjects overall satisfaction | days 1, 3,7 post-procedure
  Satisfaction ratings were classified as: very satisfied, satisfied, dissatisfied, very dissatisfied
Scab and desquamation | days 1, 3,7 post-procedure
  Record the start scab formation time, start scab removal time and complete scab removal time of subjects